CLINICAL TRIAL: NCT01355263
Title: Effect of Vitamin A Supplementation on Iron Metabolic Homeostasis of Preschool Children in Sichuan,China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu Maternal and Children's Health Care Hospital (Other)
Responsible Party: Principal Investigator, Ke Chen, headmaster, Chengdu Maternal and Children's Health Care Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20090221
Record Dates: First submitted 2011-05-09; First posted 2011-05-18 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Iron Metabolic Homeostasis
Keywords: vitamin a; preschool children; iron metabolic homeostasis; supplementation effect
MeSH Terms: interventions — Iron; Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- iron tablet, vitamin a capsule (Experimental): children in Group I received a 200,000 IU vitamin A capsule just one time initially; Group II received ferrous sulfate (element Fe 1-2 mg/kg•day) once a day for 6 months;.
  Interventions: Drug: iron and vitamin a

INTERVENTIONS:
Drug: iron and vitamin a

SUMMARY:
The investigators plan to perform a randomized, mutual-control and double-blinded cohort study to further exploit the vitamin A supplementation on iron metabolic homeostasis (including iron reserve, mobilization and absorption status in the same population) compared with solely iron and vitamin A plus iron.

ELIGIBILITY:
Inclusion Criteria:

* apparent health;
* Hb concentration>60 g/L;
* C-reaction protein (CRP)<10 mg/L;
* parental or guardian approval of participation in all aspects of the study; and
* parental/guardian agreement to avoid the additional use of vitamin and mineral supplements during the investigation.

Exclusion Criteria:

* does not match the inclusion criteria

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
hemoglobin | 6 months
hemoglobin | six months